CLINICAL TRIAL: NCT03727139
Title: AZILECT Tablets Special Drug Use-Results Survey "Survey on Long-term Safety"
Brief Title: Rasagiline Tablets Special Drug Use-Results Survey "Survey on Long-term Safety"
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Rasagiline-5001; JapicCTI-184181 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Results first posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2023-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rasagiline 1 mg: Rasagiline 1 milligram (mg), orally, once daily for up to 24 months. Participants received interventions as part of routine medical care.
  Interventions: Drug: Rasagiline

INTERVENTIONS:
Drug: Rasagiline — Rasagiline Tablets
  Other Names: AZILECT Tablets ("AZILECT" is a registered trademark of Teva Pharmaceutical Industries Ltd.)

SUMMARY:
The purpose of this survey is to evaluate the long-term safety of Rasagiline (AZILECT) in patients with Parkinson's disease in daily clinical practice and also collect efficacy information.

DETAILED DESCRIPTION:
The drug being tested in this survey is called rasagiline tablet. This tablet is being tested to treat people with Parkinson's disease.

This survey is an observational (non-interventional) study and will look at the long-term safety and efficacy of the rasagiline tablet in the routine clinical setting. The planned number of observed patients will be approximately 1000.

This multi-center observational trial will be conducted in Japan.

ELIGIBILITY:
Inclusion Criteria:

-Patients with Parkinson's disease should be surveyed.

Exclusion Criteria:

-Participants who have contraindications on package insert of rasagiline.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Parkinson's disease treated with Rasagiline 1 mg tablets as part of routine medical care.
Sampling Method: Probability Sample
Enrollment: 1021 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda Selected Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Hattori N, Kajita M, Fujimoto S, Izutsu M, Fernandez J. Safety and effectiveness of rasagiline in patients with Parkinson's disease in Japan: a post-marketing surveillance study. Expert Opin Drug Saf. 2024 Jan;23(1):79-88. doi: 10.1080/14740338.2023.2293207. Epub 2023 Dec 20. PMID 38124528
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b60294db2bf003ab49a0e

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the survey at 148 investigative sites in Japan, from 1 November 2018 to 31 October 2021.
Pre-assignment Details: Participants with a historical diagnosis of Parkinson's disease were enrolled. Participants received rasagiline as part of a routine medical care.
Period: Overall Study
Arm/Group | Rasagiline 1 mg
Started | 1021
Completed | 961
Not Completed | 60
Not completed — Protocol Violation | 60

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Arm/Group | Rasagiline 1 mg
Number analyzed (Participants) | 961
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.5 (9.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 517
  Male | 444
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — All participants were enrolled in Japan.
  Participants
    Japan | 961
Duration of Diagnosis of Parkinson's Disease [Mean (Standard Deviation); unit: Years] — Mean duration between the first diagnosis of Parkinson's disease and the start of the study was reported. Population: The number analyzed is the number of participants with data available for analysis.
  Years
    number analyzed (Participants) | 911
    (all) | 6.82 (5.405)
Healthcare Category [Count of Participants; unit: Participants] — Participants were categorized as outpatient and inpatient.
  Participants
    Outpatient | 896
    Inpatient | 65
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had No Medical Complications | 202
    Had Medical Complications | 759
Dementia [Count of Participants; unit: Participants]
  Had No Dementia | 891
  Had Dementia | 70
Height [Mean (Standard Deviation); unit: Centimeters (cm)] — Population: The number analyzed is the number of participants with data available for analysis.
  Centimeters (cm)
    number analyzed (Participants) | 712
    (all) | 157.9 (9.86)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] — Population: The number analyzed is the number of participants with data available for analysis.
  Kilograms (kg)
    number analyzed (Participants) | 722
    (all) | 54.84 (11.463)
Smoking Classification [Count of Participants; unit: Participants] — Unknown: Data could not be collected.
  Participants
    Never Smoked | 567
    Current Smoker | 19
    Ex-Smoker | 122
    Unknown | 253
Modified Hoehn & Yahr Stage [Count of Participants; unit: Participants] — Modified Hoehn & Yahr Stage represented severity for symptoms of Parkinson's disease progress. The Stage of Modified Hoehn & Yahr were assigned from Stage 0 (Asymptomatic) to Stage 5 (Wheelchair bound or bedridden unless aided (unable to walk even if aided)).
  Participants
    Stage 0 | 1
    Stage 1 | 36
    Stage 1.5 | 21
    Stage 2 | 200
    Stage 2.5 | 78
    Stage 3 | 455
    Stage 4 | 150
    Stage 5 | 20
Levodopa Use at Initiation of Treatment with the Study Drug [Count of Participants; unit: Participants]
  Not Used | 96
  Used | 865
Wearing-off Phenomenon [Count of Participants; unit: Participants] — Population: The number analyzed is the number of participants given levodopa at initiation of treatment with the study drug.
  Participants
    number analyzed (Participants) | 865
    Had No Wearing-off Phenomenon | 394
    Had Wearing-off Phenomenon | 471
Dyskinesia [Count of Participants; unit: Participants] — Population: The number analyzed is the number of participants given levodopa at initiation of treatment with the study drug.
  Participants
    number analyzed (Participants) | 865
    Had No Dyskinesia | 699
    Had Dyskinesia | 166
Unified Parkinson's Disease Rating Scale (UPDRS) Part III Total Score [Mean (Standard Deviation); unit: Scores on a Scale] — Unified Parkinson's Disease Rating Scale (UPDRS) retains the four-scale structure with a reorganization of the various subscales; (Part I) Mentation, behavior and mood (4 items), (Part II) Activities of daily living (13 items), (Part III) Motor (14 items), and (Part IV) Complications (11 items). Each item on Part III has 0-4 ratings, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe, some items were scored for 2 or more body parts. Total score range on Part III is 0-108, higher scores represent more severe symptom of Parkinson's disease (worse outcome). Population: The number analyzed is the number of participants with data available for analysis.
  Scores on a Scale
    number analyzed (Participants) | 700
    (all) | 28.5 (14.36)
Tremor Score [Mean (Standard Deviation); unit: Scores on a Scale] — UPDRS retains the four-scale structure with a reorganization of the various subscales; Part I: 4 items, Part II: 13 items, Part III: 14 items, and Part IV: 11 items. Each item on Part III has 0-4 ratings, where 0=normal, 1=slight, 2=mild, 3=moderate, and 4=severe, some items were scored for 2 or more body parts. Total score range on Part III is 0-108, higher scores represent more severe symptom of Parkinson's disease (worse outcome). Tremor score was rated 0-28 based on 2 items of the UPDRS. Higher scores represent more severe symptom of tremor. Population: The number analyzed is the number of participants with data available for analysis.
  Scores on a Scale
    number analyzed (Participants) | 716
    (all) | 3.0 (3.56)
Akinesia/Hypokinesia Score [Mean (Standard Deviation); unit: Scores on a Scale] — UPDRS retains the four-scale structure with a reorganization of the various subscales; Part I: 4 items, Part II: 13 items, Part III: 14 items, and Part IV: 11 items. Each item on Part III has 0-4 ratings, where 0=normal, 1=slight, 2=mild, 3=moderate, and 4=severe, some items were scored for 2 or more body parts. Total score range on Part III is 0-108, higher scores represent more severe symptom of Parkinson's disease (worse outcome). Akinesia/hypokinesia score was rated 0-36 based on 5 items of the UPDRS. Higher scores represent more severe symptom of akinesia/hypokinesia. Population: The number analyzed is the number of participants with data available for analysis.
  Scores on a Scale
    number analyzed (Participants) | 702
    (all) | 11.6 (6.60)
Rigidity Score [Mean (Standard Deviation); unit: Scores on a Scale] — UPDRS retains the four-scale structure with a reorganization of the various subscales; Part I: 4 items, Part II: 13 items, Part III: 14 items, and Part IV: 11 items. Each item on Part III has 0-4 ratings, where 0=normal, 1=slight, 2=mild, 3=moderate, and 4=severe, some items were scored for 2 or more body parts. Total score range on Part III is 0-108, higher scores represent more severe symptom of Parkinson's disease (worse outcome). Rigidity score was rated 0-20 based on one item of the UPDRS. Higher scores represent more severe symptom of rigidity. Population: The number analyzed is the number of participants with data available for analysis.
  Scores on a Scale
    number analyzed (Participants) | 711
    (all) | 5.9 (3.47)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had One or More Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Time Frame: 24 months
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Rasagiline 1 mg
Number analyzed (Participants) | 961
Participants | 304

2. Primary Outcome: Number of Participants Who Had One or More Adverse Drug Reactions
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. Adverse drug reaction refers to AE related to administered drug.
Time Frame: 24 months
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Rasagiline 1 mg
Number analyzed (Participants) | 961
Participants | 189

3. Secondary Outcome: Change From Baseline in the Unified Parkinson's Disease Rating Scale (UPDRS)
Description: UPDRS retains the four-scale structure with a reorganization of the various subscales; (Part I) Mentation, behavior and mood (4 items), (Part II) Activities of daily living (13 items), (Part III) Motor (14 items), and (Part IV) Complications (11 items). Each item on Part III has 0-4 ratings, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe, some items will be scored for 2 or more body parts. Total score range on Part III is 0-108, higher scores represent more severe symptom of Parkinson's disease (worse outcome).
Time Frame: Baseline, Up to Month 24 (Final Assessment Point)
Population: Efficacy assessment population, The efficacy assessment population was defined as participants who completed the survey and had efficacy data at baseline and post-baseline time points available.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Rasagiline 1 mg
Number analyzed (Participants) | 527
Scores on a scale | -2.7 (9.46)

ADVERSE EVENTS:
Time Frame: 24 months
Description: At each visit the investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to the survey treatment.
Arm/Group | Rasagiline 1 mg
All-Cause Mortality (participants affected / at risk) | 11/961
Serious Adverse Events (participants affected / at risk) | 121/961
Other Adverse Events (participants affected / at risk) | 136/961
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rasagiline 1 mg (N=961)
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 6
Pneumonia aspiration (Infections and infestations) | 4
Psoas abscess (Infections and infestations) | 1
Enteritis infectious (Infections and infestations) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Thyroid cyst (Endocrine disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 5
Delirium (Psychiatric disorders) | 2
Delusion (Psychiatric disorders) | 3
Hallucination (Psychiatric disorders) | 22
Hallucination, visual (Psychiatric disorders) | 19
Insomnia (Psychiatric disorders) | 1
Altered state of consciousness (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 4
Dementia Alzheimer's type (Nervous system disorders) | 1
Dizziness postural (Nervous system disorders) | 1
Dyskinesia (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 4
Neuroleptic malignant syndrome (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Sudden onset of sleep (Nervous system disorders) | 1
Parkinson's disease (Nervous system disorders) | 7
Aqueductal stenosis (Nervous system disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure chronic (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Aortic dissection (Vascular disorders) | 1
Blood pressure fluctuation (Vascular disorders) | 2
Hypertension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 6
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Rectal stenosis (Gastrointestinal disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Congestive hepatopathy (Hepatobiliary disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1
Azotaemia (Renal and urinary disorders) | 1
Neurogenic bladder (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Death (General disorders) | 1 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
Drowning (General disorders) | 1
Sudden death (General disorders) | 2 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
Multiple organ dysfunction syndrome (General disorders) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Fibrin D dimer increased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Fall (Injury, poisoning and procedural complications) | 5
Femoral neck fracture (Injury, poisoning and procedural complications) | 5
Femur fracture (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 1
Patella fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 6
Subdural haematoma (Injury, poisoning and procedural complications) | 3
Pelvic fracture (Injury, poisoning and procedural complications) | 2
Heat illness (Injury, poisoning and procedural complications) | 1
Hospitalisation (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rasagiline 1 mg (N=961)
Dizziness (Nervous system disorders) | 14
Dyskinesia (Nervous system disorders) | 40
Somnolence (Nervous system disorders) | 15
Orthostatic hypotension (Vascular disorders) | 24
Nausea (Gastrointestinal disorders) | 15
Fall (Injury, poisoning and procedural complications) | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT03727139/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT03727139/SAP_001.pdf